CLINICAL TRIAL: NCT05896683
Title: A Phase 1, Open-label, Randomized, 2-Part, 2-Way Crossover Study in Healthy Adult Participants to Assess the Relative Bioavailability of Tablet Formulations of Lazertinib (JNJ-73841937)
Brief Title: A Study of Lazertinib (JNJ-73841937) Tablet in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: CR109314; 73841937NSC1010 (Other: Janssen Research & Development, LLC); 2022-502814-99-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2023-06-01; First posted 2023-06-09 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — lazertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part 1: Sequence AB (Experimental): Participants will receive intervention A (lazertinib reference formulation) on Day 1 of intervention period 1. After washout period of 14 to 21 days, participants will receive intervention B (lazertinib test formulation) on Day 1 of intervention period 2.
  Interventions: Drug: Lazertinib
- Part 1: Sequence BA (Experimental): Participants will receive intervention B (lazertinib test formulation) on Day 1 of intervention period 1. After washout period of 14 to 21 days, participants will receive intervention A (lazertinib reference formulation) on Day 1 of intervention period 2.
  Interventions: Drug: Lazertinib
- Part 2: Sequence CD (Experimental): Participants will receive Intervention C (lazertinib reference formulation) on Day 1 of intervention period 1. After washout period of 14 to 21 days, participants will receive intervention D (lazertinib test formulation) on Day 1 of intervention period 2.
  Interventions: Drug: Lazertinib
- Part 2: Sequence DC (Experimental): Participants will receive intervention D (lazertinib test formulation) on Day 1 of intervention period 1. After washout period of 14 to 21 days, participants will receive intervention C (lazertinib reference formulation) on Day 1 of intervention period 2.
  Interventions: Drug: Lazertinib

INTERVENTIONS:
Drug: Lazertinib — Lazertinib will be administered orally.
  Other Names: JNJ-73841937

SUMMARY:
The purpose of this study is to assess the extent of availability of drug to the body of four different lazertinib tablet formulations at a single oral dose under fasted conditions in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical examination, medical history (at screening only), vital signs, and 12-lead electrocardiogram (ECG) performed at screening and at admission to the study site in Intervention Period 1
* Body weight not less than 50.0 kilograms (kgs) and body mass index (BMI, weight/height^2) within the range 19.0-30.0 kg/m^2 (inclusive) at screening
* All female participants must have a negative highly sensitive serum beta-human chorionic gonadotropin (beta-HCG) test at screening and a negative urine pregnancy test on Day -1 of Intervention Period 1
* A male participant must agree not to donate sperm for the purpose of reproduction during the study and for a minimum of 6 months after receiving the last dose of study intervention
* Must sign an ICF indicating that the participant understands the purpose of, and procedures required for, the study and is willing to participate in the study

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease and interstitial lung disease, diabetes mellitus (with the exception of history of gestational diabetes), hepatic insufficiency, inflammation bowel disease/Crohn's disease, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* History of stomach or intestinal surgery or resection, including cholecystectomy, that would potentially alter absorption or excretion of orally administered drugs
* History of malignancy within 5 years before screening
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for paracetamol, ibuprofen, and stable hormone replacement therapy (in postmenopausal female participants only) within 14 days before the first dose of study intervention is scheduled until completion of the study
* History of human immunodeficiency virus (HIV) antibody positive, or tests positive for HIV at screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Part 1: Maximum Observed Plasma Concentration (Cmax) of Lazertinib | Pre dose up to 168 hours post dose on Day 1
  Cmax is defined as maximum observed plasma concentration of lazertinib.
Part 2: Maximum Observed Plasma Concentration (Cmax) of Lazertinib | Pre dose up to 168 hours post dose on Day 1
  Cmax is defined as maximum observed plasma concentration of lazertinib.
Part 1: Area Under the Plasma Concentration-time Curve from Time 0 to 72 Hours (h) (AUC[0-72h]) of Lazertinib | Pre dose up to 72 hours post dose on Day 1
  AUC(0-72h) is the area under the plasma concentration-time curve from time 0 to 72 hours.
Part 2: Area Under the Plasma Concentration-time Curve from Time 0 to 72h (AUC[0-72h]) of Lazertinib | Pre dose up to 72 hours post dose on Day 1
  AUC(0-72h) is the area under the plasma concentration-time curve from time 0 to 72 hours.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Up to 8 Weeks
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention.
Number of Participants With Serious Adverse Events (SAEs) | Up to 8 Weeks
  A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Number of Participants With AEs by Severity | Up to 8 Weeks
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. Number of participants with AEs by severity will be reported. Severity will be graded according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from grade 1 to 5, where Grade 1= mild, Grade 2= moderate, Grade 3= severe, Grade 4= life-threatening and Grade 5= death related to adverse event.
Number of Participants With Change From Baseline in Clinical Laboratory Test Values | Up to 8 Weeks
  Number of participants with change from baseline in clinical laboratory test values (including hematology and serum chemistry) will be reported.
Number of Participants With Change From Baseline in 12-lead Electrocardiograms (ECGs) | Up to 8 Weeks
  Number of participants with change from baseline in 12-lead ECGs will be reported.
Number of Participants With Change From Baseline in Vital Signs | Up to 8 Weeks
  Number of participants with change from baselines in vital signs (including temperature [oral], pulse rate, and blood pressure) will be reported.
Number of Participants With Change From Baseline in Physical Examination | Up to 8 Weeks
  Number of participants with change from baseline in physical examination (including height and body weight) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- SGS Belgium NV, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency